CLINICAL TRIAL: NCT05727059
Title: Early Feasibility Study (EFS) of the Magenta Elevate™ Percutaneous Left Ventricular Assist Device (pLVAD) System in Patients Undergoing Non-emergent, High-risk Percutaneous Coronary Interventions
Brief Title: Magenta Elevate™ EFS in High-Risk PCI Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Magenta Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DRD00417
Record Dates: First submitted 2023-01-25; First posted 2023-02-14 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: High-risk Percutaneous Coronary Intervention
Keywords: HRPCI; High-risk percutaneous coronary intervention; Circulatory support; Left ventricular unloading

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- HR-PCI patients (Experimental): Patients undergoing non-emergent, high-risk percutaneous coronary interventions
  Interventions: Device: The Elevate™ System

INTERVENTIONS:
Device: The Elevate™ System — The Magenta Elevate™ is a temporary (≤ 6 hours) ventricular support device indicated for use during high-risk percutaneous coronary interventions (PCI) performed electively or urgently in hemodynamically stable patients, with severe coronary artery disease.

SUMMARY:
The Elevate™ EFS study is designed to evaluate the safety and feasibility of the Magenta Elevate™ percutaneous Left Ventricular Assist Device (pLVAD) System in patients undergoing non-emergent, high-risk percutaneous coronary interventions.

DETAILED DESCRIPTION:
The Elevate™ EFS is planned as a prospective, single-arm, interventional multi-center study enrolling up to 20 subjects.

The Magenta Elevate™ Pump is a catheter-mounted, self-expanding and retrievable pump, designed to unload the left ventricle by actively transporting blood from the left ventricle into the ascending aorta.

The Magenta Elevate™ is a temporary (≤ 6 hours) ventricular support device indicated for use during high-risk percutaneous coronary interventions (PCI) performed electively or urgently in hemodynamically stable patients, with severe coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

1. Non-emergent, percutaneous coronary intervention is planned in at least one stenotic lesion of a native coronary artery or bypass graft (de novo or restenosis).
2. Ejection fraction of ≤ 50% and at least one of the following:

   1. Intervention on an unprotected left main coronary artery
   2. Intervention on a last patent coronary conduit
   3. Three-vessel disease (in case of left coronary artery dominance, the combination of a left anterior descending artery (LAD) lesion and a proximal left circumflex artery (LCX) lesion qualifies as three-vessel disease).
3. A heart team that includes a cardiac surgeon has determined that high-risk PCI is the appropriate therapeutic option.
4. Subject signed informed consent.

Exclusion Criteria:

1. Subject age < 18 or ≥ 85 years.
2. Cardiogenic shock (systolic blood pressure < 90 mmHg with evidence of end organ hypoperfusion, such as cool extremities or urine < 30 mL/hour); acutely decompensated pre-existing chronic heart failure; any use of inotropic or vasopressor in the previous 48 hours; or any use of mechanical circulatory support or an extracorporeal membrane oxygenation device within 14 days.
3. Hypertrophic cardiomyopathy, restrictive cardiomyopathy, or constrictive pericarditis
4. Evidence of left ventricular thrombus.
5. Previous aortic valve replacement or repair or a heart-constrictive device.
6. Aortic stenosis
7. Aortic regurgitation (≥ 2+ on a 4-grade scale by Transthoracic Echocardiography).
8. Aortic pathology, such as aortic aneurysms, dissection, extreme tortuosity, calcifications, or prior aortic surgery, that could pose undue additional risk to the placement of a pLVAD device.
9. Left ventricle rupture.
10. Cardiac tamponade.
11. Subject is scheduled for a staged PCI within 90 days of the index procedure
12. Subject has any condition or scheduled surgery that will require discontinuation of the antiplatelet and/or anticoagulant therapy within 90 days of the index procedure.
13. Chronic renal dysfunction (eGFR <30 mL/min/1.73 m²) and patients requiring renal replacement therapy with dialysis.
14. Known or suspected coagulopathy or abnormal coagulation parameters (defined as platelet count ≤ 100,000 or spontaneous INR ≥ 1.5 or known fibrinogen ≤ 1.5 g/L).
15. Infection of the proposed procedural access site or suspected systemic active infection, including any fever.
16. Active COVID-19 infection.
17. Stroke or transient ischemic attack within 6 months of enrollment.
18. Subject participation in another investigational drug or device trial (with the exception of post-market registries and observational studies, subject to Sponsor review and approval).
19. Female subjects who are pregnant or breast-feeding.
20. Any non-cardiac condition with a life expectancy <24 months
21. Subject has other medical, social, or psychological problems that, in the opinion of the Investigator, compromises the subject's ability to provide written informed consent and/or to comply with study procedures.
22. Subject belongs to a vulnerable population defined as individuals with mental disability, persons in nursing homes, children, impoverished persons, homeless persons, nomads, refugees, and those permanently incapable of providing informed consent. Vulnerable populations also may include members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, employees of the Sponsor, members of the armed forces, and persons kept in detention.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
Rate of Major Device-Related Adverse Events (MDRAE) | From device delivery through device removal (up to 6 hours)
  The rate of Elevate™ related Serious Adverse Events
Rate of successful initiation and maintenance of hemodynamic support without Severe Hypotension | From device delivery through device removal (up to 6 hours)
  Rate of successful initiation and maintenance of Elevate™ hemodynamic support without Severe Hypotension

SECONDARY OUTCOMES:
Rate of Elevate™ Technical Success | From device delivery through device removal (up to 6 hours)
  The rate of complete Elevate™ Pump delivery procedures, including operation of the Pump without Device Malfunction and successful retrieval of the Pump
Rate of Elevate™ Procedural Success | From device delivery through device removal (up to 6 hours)
  The rate of Elevate™ Technical Success without Severe Hypotension
Rate of Major Device-Related Adverse Events (MDRAE) | From device removal through hospital discharge (assessed up to 30 days)
  The rate of Elevate™ related Serious Adverse Events
Rate of Major Device-Related Adverse Events (MDRAE) | From hospital discharge through 30-days post device removal
  The rate of Elevate™ related Serious Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Zohar Bronshtine, Study Director — Magenta Medical Ltd.
Locations (2):
- United States (2):
  - Mount Sinai Hospital, New York, New York
  - New York-Presbyterian Hospital/Columbia University Irving Medical Center, New York, New York